CLINICAL TRIAL: NCT03256136
Title: A Phase II Study of Nivolumab in Combination With Carboplatin and Pemetrexed, or Nivolumab in Combination With Ipilimumab, in Patients With Advanced, EGFR-mutant or ALK-rearranged, Non-Small Cell Lung Cancer
Brief Title: Nivolumab in Combination With Chemotherapy, or Nivolumab in Combination With Ipilimumab, in Advanced EGFR-Mutant or ALK-Rearranged NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Alice Shaw, Director, Center for Thoracic Cancers, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-011
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Nivolumab; Pemetrexed; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nivolumab Plus Ipilimumab EGFR (Experimental): Nivolumab administered intravenously every 2 weeks Ipilimumab administered intravenously every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivolumab Plus Ipilimumab ALK (Experimental): Nivolumab administered intravenously every 2 weeks Ipilimumab administered intravenously every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Nivolumab + Carboplatin + Pemetrexed with EGFR Chemo naive (Experimental): Nivolumab administered intravenously every 3 weeks Carboplatin administered intravenously every 3 weeks Pemetrexed administered intravenously every 3 weeks
  Interventions: Drug: Carboplatin; Drug: Nivolumab; Drug: pemetrexed
- Nivolumab + Carboplatin + Pemetrexed ALK Chemo naive (Experimental): Nivolumab administered intravenously every 3 weeks Carboplatin administered intravenously every 3 weeks Pemetrexed administered intravenously every 3 weeks
  Interventions: Drug: Carboplatin; Drug: Nivolumab; Drug: pemetrexed

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy
  Other Names: Paraplatin
  Arms: Nivolumab + Carboplatin + Pemetrexed ALK Chemo naive; Nivolumab + Carboplatin + Pemetrexed with EGFR Chemo naive
Drug: Nivolumab — will allow the body's immune system to work against tumor cells
  Other Names: Opdivo
Drug: pemetrexed — Chemo therapy
  Other Names: Alimta
  Arms: Nivolumab + Carboplatin + Pemetrexed ALK Chemo naive; Nivolumab + Carboplatin + Pemetrexed with EGFR Chemo naive
Drug: Ipilimumab — will allow the body's immune system to work against tumor cells
  Other Names: Yervoy
  Arms: Nivolumab Plus Ipilimumab ALK; Nivolumab Plus Ipilimumab EGFR

SUMMARY:
This research study is studying a drug intervention as a possible treatment for lung cancer.

The drugs involved in this study are:

* Nivolumab
* Carboplatin
* Pemetrexed
* Ipilimumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease.

The FDA (the U.S. Food and Drug Administration) has approved Nivolumab as a treatment for other types of cancers including lung cancer. However, the combination of Nivolumab with other drugs (such as those being tested in this study) has not been approved by the FDA as a treatment for this type of lung cancer.

The purpose of this study is to test the effectiveness (how well the drug works), safety, and tolerability of the drug Nivolumab in combination with standard of care chemotherapies, or in combination with Ipilimumab. Nivolumab and Ipilimumab are antibodies (a type of human protein) that are being tested to see if they will allow the body's immune system to work against tumor cells. This study is being done to see if Nivolumab and Ipilimumab, or Nivolumab and chemotherapy drugs (Carboplatin and Pemetrexed), are more effective against cancer when administered together.

These drugs are given as infusions. They are designed to "boost" the immune system's ability to suppress or kill cancer cells that are foreign to the human body.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced (stage IIIB or IV) non-small-cell lung cancer (NSCLC).

  * ALK-rearranged NSCLC: ALK rearrangement as assessed by ALK FISH, IHC, or next-generation sequencing (NGS). For ALK FISH, rearrangements must be detected in >15% of tumor cells.
  * EGFR-mutant NSCLC: EGFR activating gene mutation (e.g., L858R, exon 19 deletion) as well as a T790M mutation per local testing.
* Presence of at least one measurable lesion as defined by RECIST v1.1. A previously irradiated site lesion may only be counted as a target lesion if there is clear sign of progression since the completion of irradiation.
* Prior treatment with appropriate tyrosine kinase inhibitors (TKIs) as follows:

  * ALK-positive NSCLC (cohorts B and D): Participants must have progressed on or after 1 or more next-generation ALK-TKI(s).
  * EGFR-mutant NSCLC (cohorts A and C): Participants must have progressed on or after 1 or more third-generation, T790M mutant-selective EGFR-TKI(s).
* Prior systemic chemotherapy requirements are as follows:

  * Nivolumab plus carboplatin and pemetrexed arms (cohorts A and B): NO prior systemic chemotherapy is allowed. NOTE: Prior adjuvant or neoadjuvant chemotherapy is allowed if received more than 12 months prior to the study.
  * Nivolumab plus ipilimumab arms (cohorts C and D): Participants must have received a platinum-based combination chemotherapy for their advanced lung cancer and either progressed on/after this chemotherapy or are intolerant. Only ONE line of chemotherapy is allowed. NOTE: Prior adjuvant or neoadjuvant chemotherapy does not count as an additional line of chemotherapy if received more than 12 months prior to the study.
* Tumor tissue sample is required following the participant's last line of systemic therapy (TKI or chemotherapy). Tissue sample may be fresh (core needle, excisional, or incisional biopsy), or archival if obtained within 6 months prior to enrollment. There can have been no systemic therapy administered after the sample was obtained. If a tissue sample is available but it has been > 6 months and there has been no intervening therapy, the Principal Investigator may approve the sample after discussion. PD-L1 IHC testing will be performed on the tumor tissue, but positivity on the PD-L1 IHC testing is not required to enroll in the study.
* Clinically asymptomatic and stable central nervous system (CNS) metastases are allowed (including untreated CNS metastases) if they have not required increasing doses of steroids or stable doses equivalent to prednisone > 10 mg daily within 2 weeks prior to study entry for CNS symptoms.
* Prior palliative radiotherapy must have been completed at least 2 weeks prior to study entry.
* Subjects must have been off any prior systemic anti-cancer treatment (including TKIs) for at least 5 half-lives of that drug.
* Age ≥ 18 years old.
* ECOG performance status of 0 or 1.
* Life expectancy ≥ 12 weeks.
* Screening laboratory values must meet the following criteria:

  * WBC ≥ 2.0 x 109/L
  * Neutrophils ≥ 1.5 x 109/L
  * Platelet ≥ 100 x 109/L
  * Hemoglobin ≥ 9/dL
  * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance using Cockcroft-Gault formula ≥ 50 mL/min

    * Female CrCl = (140-age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
    * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
  * Total bilirubin ≤ 1.5 x ULN (except in patients with Gilbert's syndrome who may have total bilirubin < 3.0 mg/dL)
  * AST and ALT ≤ 3.0 x ULN (or ≤ 5.0 x ULN if liver metastases are present)
* Females of child-bearing potential (defined as a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy or has not been naturally post-menopausal for at least 24 consecutive months) must:

  * Have a negative serum or urine pregnancy test obtained within 24 hours prior to starting the investigational drug.
  * Not be breastfeeding.
  * Agree to use, and be able to comply with, highly effective contraception (failure rate less than 1% per year) without interruption while on study treatment plus 5 half-lives of nivolumab (half-life up to 25 days) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post treatment completion. Complete abstinence is acceptable if it is in line with the preferred and usual lifestyle of the patient. Period abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal implants, established and proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods from the options of diaphragm, cervical cap, vaginal sponge, and condom, or progesterone-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
* Male subjects agree to remain abstinent or use a condom plus an additional contraceptive method that result in a failure rate of <1% per year during sexual contact with a female of childbearing potential while participating in the study, during dose interruptions, and for 31 weeks following the last dose of the study treatment, even if he has undergone a successful vasectomy. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable.
* Subject has the ability to understand and provide signed informed consent.
* Subject has the willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Subjects previously treated with T cell immune-modulating antibodies, including anti-CTLA-4, anti-PD-1 and/or anti-PD-L1 agents.
* Subjects with symptomatic brain metastases, carcinomatous meningitis, spinal cord compression, or intractable back pain due to compression of destructive mass.
* Subjects with active, known, or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization (unless used to treat investigational drug-related adverse events). Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Subjects with interstitial lung disease or interstitial pneumonitis that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days prior to screening. No major surgery, other than diagnostic surgery, is allowed within 4 weeks prior to treatment in the study.
* Co-administration of anti-cancer therapies other than those administered in the study.
* Subjects with other active malignancy requiring concurrent intervention.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). HIV-positive participants are ineligible because these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy, and because there is the potential for pharmacokinetic interactions with combination antiretroviral therapy and study drugs.
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Subjects with ≥ grade 2 peripheral neuropathy at enrollment per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
* Pregnant or lactating women. Pregnant women are excluded from this study because the study drugs (i.e., nivolumab, ipilimumab, carboplatin, and pemetrexed) have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued.
* Subjects currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug.
* History of allergy or hypersensitivity to any study drugs or their excipients.
* Any known clinically significant concomitant medical condition, laboratory abnormality, or psychiatric illness that, in the investigator's opinion, would prevent the subject from participating in the study, pose an unacceptable risk to the patient in this study, or interfere with the interpretation of safety results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shaw, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts general Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Started | 3 | 1 | 4 | 1
Completed | 3 | 1 | 4 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive | Total
Number analyzed (Participants) | 3 | 1 | 4 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 1 | 5
  >=65 years | 2 | 0 | 2 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 4
  Male | 1 | 0 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 2 | 1 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4 | 1 | 9
Treatment Regimen Received [Count of Participants; unit: Participants] | 3 | 1 | 4 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Presented in Numbers of Participants
Description: Complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Number analyzed (Participants) | 3 | 1 | 4 | 1
Participants | 0 | 0 | 1 | 1

2. Secondary Outcome: Disease Control Rate (DCR), Presented in Numbers of Participants
Description: The number of patients that achieved either complete response (CR), partial response (PR), or stable disease (SD) per RECIST version 1.1
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Number analyzed (Participants) | 3 | 1 | 4 | 1
Participants | 0 | 0 | 3 | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from initiation of the study drugs to progression or death, whichever occurs first. Disease progression was assessed via RECIST 1.1
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study(this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progression).
  Confidence Intervals (CIs) were calculated using the Kaplan Meier (KM) method
Time Frame: From the start of treatment until disease progression or death due to any cause, up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Number analyzed (Participants) | 3 | 1 | 4 | 1
months | 1.3 [0.6 to 1.4] | 0.7 [NA to NA] — confidence interval is not defined due to an insufficient number of events | 4.65 [1.2 to 8.4] | 2.8 [NA to NA] — confidence interval is not defined due to an insufficient number of events

4. Secondary Outcome: Overall Survival (OS)
Description: Time from initiation of the study drugs to date of death due to any cause. CIs are the KM estimate CIs.
Time Frame: From the start of treatment until death due to any cause, up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Number analyzed (Participants) | 3 | 1 | 4 | 1
months | 22.3 [2.6 to 23.7] | 7.6 [NA to NA] — confidence interval is not defined due to an insufficient number of events | 7.75 [2.1 to 16.2] | 15.9 [NA to NA] — confidence interval is not defined due to an insufficient number of events

5. Secondary Outcome: Duration Of Response
Description: Time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause, whichever occurs first
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study(this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progression).
Time Frame: From the first documented response until disease progression or death, up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
Number analyzed (Participants) | 3 | 1 | 4 | 1
months | NA [NA to NA] — no objective responses in this cohort | NA [NA to NA] — no objective responses in this cohort | 0.9 [NA to NA] — confidence interval is not defined due to an insufficient number of events | 1.4 [NA to NA] — confidence interval is not defined due to an insufficient number of events

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, up to approximately 2 years
Arm/Group | Nivolumab Plus Ipilimumab EGFR | Nivolumab Plus Ipilimumab ALK | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/1 | 2/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/1 | 3/4 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 0/1 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Plus Ipilimumab EGFR (N=3) | Nivolumab Plus Ipilimumab ALK (N=1) | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive (N=4) | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive (N=1)
Blood bilirubin increase (Investigations) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutrophil count decrease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Plus Ipilimumab EGFR (N=3) | Nivolumab Plus Ipilimumab ALK (N=1) | Nivolumab + Carboplatin + Pemetrexed With EGFR Chemo Naive (N=4) | Nivolumab + Carboplatin + Pemetrexed ALK Chemo Naive (N=1)
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 4 | 0
Pain (General disorders) | 1 | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 2 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0
General disorders, other - Tick bite (General disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Nervous system disorders, other - numbness to chin and extremities (Nervous system disorders) | 0 | 0 | 1 | 0
Gum infection (Infections and infestations) | 0 | 0 | 1 | 0
Platelet count decreased (Infections and infestations) | 0 | 0 | 2 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Eye disorders - other: red vision (Eye disorders) | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0
Lymphocyte decreased (Investigations) | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03256136/Prot_SAP_000.pdf